CLINICAL TRIAL: NCT07371585
Title: Patient-Centered Study of Trastuzumab Deruxtecan (T-DXd) in First-Line HER2-Positive Metastatic Breast Cancer With Proactive Toxicity Management Reflecting Real-World Clinical Practice
Brief Title: Trastuzumab Deruxtecan in First-Line HER2-Positive Metastatic Breast Cancer With Proactive Toxicity Management
Acronym: TOP-REAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Collaborators: Westdeutsche Studiengruppe GmbH (WSG) (Unknown); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-2402; 2025-521805-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-30; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Stage IV
Keywords: Trastuzumab deruxtecan; digital health tools; first line; proactive toxicity management
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-DXd + pertuzumab + digital health tools (Experimental): Trastuzumab Deruxtecan (T-DXd) in combination with pertuzumab, together with the use of digital health tools
  Interventions: Device: Digital Health Tools; Drug: T-DXd; Drug: Pertuzumab

INTERVENTIONS:
Device: Digital Health Tools — Patients will be followed via digital health tools for proactive toxicity management, which consist of one mobile app and two devices: (1) CANKADO/Resilience app (depending on the country and site) accessed through the patient's phone; (2) A pulse oximeter that together with the digital health mobile app will allow self-tracking of vital parameters such as oxygen saturation and heart rate, potentially facilitating early ILD detection; and (3) A smartwatch to collect patient granular data. All three digital health tools/items are CE-marked medical devices, where relevant, used exclusively within their approved intended purpose, and not subject to any investigation of safety or performance within this study.
  Other Names: CANKADO; Resilience; Pulse oximeter; Smartwatch
Drug: T-DXd — T-DXd at 5.4 mg/kg will be administered as IV infusion q3w.
  Other Names: Trastuzumab deruxtecan + Pertuzumab; Pertuzumab
Drug: Pertuzumab — Pertuzumab will be administered at a loading dose of 840 mg on Day 1 of Cycle 1, followed by 420 mg in subsequent cycles, administered as IV q3w.

SUMMARY:
This is an open-label, single arm, non-randomized, multicenter, phase 2 study assessing the efficacy and safety of T-DXd as first-line treatment in HER2-positive advanced/metastatic BC patients (N=300). The study integrates digital health tools for proactive toxicity management and potentially facilitate early detection of ILD/pneumonitis.

DETAILED DESCRIPTION:
*Study Population*

The study will enroll male or pre/post-menopausal women aged ≥ 18 years with locally advanced or metastatic HER2-positive (IHC 3+ or ISH+, by local testing) BC who have not received prior chemotherapy or HER2-targeted therapy for advanced/metastatic disease. Eligible patients should have evaluable disease (measurable and not measurable) as defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Patients with active and treated CNS metastases not requiring immediate local therapy are eligible.

*Study Interventions *

Patients meeting all eligibility criteria will receive T-DXd at 5.4 mg/kg administered as IV infusion q3w in combination with pertuzumab at a loading dose of 840 mg on Day 1 of Cycle 1, followed by 420 mg in subsequent cycles, administered as IV q3w. Treatment will be administered continuously until RECIST 1.1-defined progressive disease, unacceptable toxicity, investigator's decision, withdrawal of consent, or other reasons described in the protocol. T-DXd rechallenge will be allowed for patients who discontinued T-DXd for reasons other than progressive disease, grade ≥2 ILD or any toxicity requiring permanent discontinuation per T-DXd SmPC and/or protocol-defined management guidelines, and who have progressed to maintenance treatment. Standard endocrine therapy (aromatase inhibitor, fulvestrant or tamoxifen) administered concurrently with the study treatment (from C1D1) is allowed for patients with HR-positive tumors, as per local practice. For men and premenopausal women, LHRH agonist is allowed as per local practice.

Patients will be followed via digital health tools. These consist of one mobile app and two devices:

* Digital health mobile app (CANKADO or Resilience depending on the country and site [used in accordance with respective CE markings]) accessed through the patient's phone and offering:

  * Remote (Resilience PRO) or automated (CANKADO PRO-react) patient monitoring through electronic patient-reported outcomes (ePROs).
  * Comprehensive educational content with a focus on managing study treatment-related toxicities.
  * Optional self-management programs to support patient autonomy, including cognitive behavioral therapy for fatigue, adapted physical activity, and meditation (Resilience only).
* A pulse oximeter that together with the digital health mobile app will allow self-tracking of vital parameters such as oxygen saturation and heart rate, potentially facilitating early ILD detection.
* A smartwatch to collect patient granular data.

*Study Assessments *

Imaging will be performed prior to day 1 of treatment and target and non-target lesions will be identified as per RECIST v.1.1. Tumor assessments will be performed every 9 weeks for the first 12 months from start of treatment and then every 12 weeks until disease progression, withdrawal of consent, death, or the end of the study, whichever occurs the first. Tumor assessments will be performed on the specified schedule regardless of treatment delays. Tumor response will be assessed as per RECIST v.1.1.

A Formalin-Fixed Paraffin Embedded (FFPE) specimen from metastatic disease (preferably) with adequate quantity and quality of tumor tissue must be provided (tumor block) prior to treatment. Samples will be tested to confirm quality at the central lab prior to enrollment. Remaining tissue will be kept at the central lab for retrospective HER2 central confirmation and additional biomarkers of response. A tumor biopsy will be also performed at disease progression. Blood samples (for biomarkers) will be collected at C1D1, C2D1 and at disease progression for exploratory objectives.

Patients that discontinue for reasons other than progressive disease, ILD/pneumonitis ≥ Grade 2 or any toxicity requiring permanent discontinuation per T-DXd SmPC and/or protocol-defined management guidelines, will go through a structured interview at the moment of T-DXd discontinuation. This structured interview will collect information from both the healthcare professional and the patient at that time to understand the main reasons for T-DXd discontinuation and if the patient is deemed "suitable" or "not suitable" for T-DXd rechallenge. This interview will also be conducted before treatment restart. Blood samples will be collected at C1D1, C2D1 and disease progression during T-DXd rechallenge.

A blood sample will be collected from each patient at C2D1 to obtain germline DNA for Pharmacogenomic analyses.

PRO instruments will be completed by patients to evaluate the treatment impact from the patient's perspective.

All patients will be closely monitored for adverse events (AEs) throughout the study. The incidence, nature, and severity of AEs and laboratory abnormalities will be graded per the NCI CTCAE v.5.0. Laboratory safety assessments will include the regular monitoring of hematology, serum chemistry, oxygen saturation and pregnancy test. Oxygen saturation and heart rate will also be monitored once a day by the digital health tools. Primary prophylaxis for the prevention of nausea and vomiting with a combination of three (3) antiemetic agents (e.g., dexamethasone with either a 5 HT3 receptor antagonist and/or an NK1 receptor antagonist, as well as other medicinal products as indicated) is mandatory.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the nature of the study and to voluntarily provide written informed consent prior to any trial-specific screening procedures and has sufficient cognitive capacity to comply with study requirements, including the use of digital health tools and devices.
2. Male/female patients who are at least 18 years of age on the day of signing informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Histologically or cytologically locally confirmed HR+/HER2+ or HR-/HER2+ BC with evidence of locally advanced disease, not amenable to resection or radiation therapy with curative intent, or metastatic disease:

   1. HER2-positivity confirmed in a tumor sample obtained in the metastatic setting, defined as either IHC 3+ or in situ hybridization positive (ISH+) by local laboratory assessment as per the most recent American Society of Clinical Oncology (ASCO)-College of American Pathologists Guideline (CAP) guideline. The most recent test result prior screening period will be used to confirm eligibility.
   2. Documented HR (ER and/or PR) positivity or negativity, confirmed by local laboratory assessment in a tumor sample obtained in the metastatic setting. ER and/or PR positivity is defined as >1% of cells expressing HR via IHC analysis as per most recent ASCO-CAP guideline. The most recent test result prior screening period will be used to confirm eligibility.
5. No prior chemotherapy or HER2-targeted therapy for advanced or mBC (1 prior line of endocrine therapy is allowed for mBC). Participants who have received chemotherapy or HER2-targeted therapy in the neoadjuvant or adjuvant setting at any time are eligible.

   Note: Patients that received an antibody-drug conjugate containing an exatecan derivative (topoisomerase I inhibitor) in the adjuvant setting, must have a disease-free interval of ≥12 months since the last dose.
6. Evaluable disease as defined by RECIST v1.1.

   Note: Previously irradiated lesions can be considered as measurable disease only if disease progression has been unequivocally documented at that site since radiation.
7. Adequate FFPE tumor tissue sample available from the metastatic setting (preferably) for retrospective HER2 central analysis confirmed by central laboratory. An adequate sample of tumor tissue must be provided from either a newly acquired biopsy from a region that has not been previously irradiated or the most recent archival sample.
8. Patients with Brain Metastases (BM): Eligible if either previously untreated or previously treated BM, provided there is no clinical indication for immediate local therapy. For untreated BM, lesions must be ≤2.0 cm in largest diameter; lesions >2.0 cm require discussion with and approval from the Medical Monitor. Patients must not require >3 mg/day of dexamethasone (or equivalent corticosteroid) for symptom control. If receiving anticonvulsants, the regimen must be stable for ≥14 days prior to first dose. A washout period prior enrollment of ≥3 weeks since stereotactic radiosurgery or gamma knife, whole-brain radiotherapy, or radiotherapy or surgery for spinal cord compression is required.

   Note: Patients with leptomeningeal disease may be eligible after discussion with the Medical Monitor.
9. Adequate hematologic and end-organ function, defined by the following laboratory results (see protocol)
10. LVEF ≥ 50% within 28 days before Cycle 1 Day 1.
11. Life expectancy of ≥ 12 weeks at screening.
12. Adequate treatment washout period before first dose of study intervention, defined as (see protocol)
13. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified highly effective method of contraception.
14. Access to a smartphone with internet connection that allows them to carry out the required assessments at the specified timepoints and with the following characteristics:

    * Resilience PRO: Android 8.0 (or newer) OR iOS 15.0 (or newer)
    * Cankado PRO-React: Android 13.0 (or newer) OR iOS 17.0 (or newer)
15. Only applicable in France: patients affiliated to the social security system.

Exclusion Criteria:

1. Patients with HER2-negative disease.
2. Subjects who, in the opinion of the investigator, are unable to comply with the protocol requirements or who have any comorbidity or condition that may hinder study follow-up, response evaluation, or the informed consent process, including inability to read and understand the local language of the study site sufficiently to interact effectively with study materials and tools (including digital applications).

   Note: Other languages for app-based questionnaires may be provided upon patient request and based on availability of such questionnaires and tools.
3. History of other primary malignancy unless treated with curative intent with no evidence of active disease within 3 years before the first dose of study treatment and of low potential risk for recurrence. Exceptions include: basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy, adequately resected non-melanoma skin cancer, in situ cancer of the cervix, curatively treated ductal carcinoma in situ (DCIS), contralateral breast cancer, Stage 1, grade 1 endometrial carcinoma or other solid malignant tumors with an expected curative outcome after Medical Monitor approval.
4. Persistent toxicities that the investigator deems related to previous anti-cancer therapy (excluding alopecia), not yet resolved to grade ≤ 1 or baseline. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study treatment may be included (e.g., hearing loss). Participants with stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to enrollment and managed with standard of care treatment) may be eligible per the discretion of the investigator (e.g., Grade 2 chemotherapy-induced neuropathy).
5. Untreated spinal cord compression
6. History of significant cardiovascular disease, defined as:

   * New York Heart Association Class III or greater congestive heart failure or known left ventricular ejection fraction of < 50%.
   * Participants with a medical history of myocardial infarction within 6 months before enrollment or symptomatic CHF (NYHA Class II to IV). Participants with troponin levels above upper limit of normal (ULN) at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out myocardial infarction.
   * History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation (Mean resting corrected QTcF interval >470ms (females) or >450msec (males)). Note: Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted upon discussion with the Medical Monitor.
7. History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening. Patients with a history of grade 1 drug-induced ILD/pneumonitis, who are now fully recovered, must be discussed with the Medical Monitor for approval.
8. Meets one of the following lung criteria:

   * Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within 3 months of study enrollment, prior pneumonectomy (complete), severe asthma, severe chronic obstructive pulmonary disorder (COPD), restrictive lung disease, pleural effusion, post COVID-19 pulmonary fibrosis, etc,).
   * Any autoimmune, connective tissue or inflammatory disorders (eg, rheumatoid arthritis, Sjogren's, sarcoidosis, etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the electronic Case Report Form (eCRF) for participants who are included in the study.
9. Received a live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of study treatment.

   Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of study treatment.
10. Active serious infection requiring IV antibiotics, antivirals, or antifungals.
11. Active HIV, HBV (defined as having a positive HbsAg test) or HCV.

    1. Participants with a known history of human immunodeficiency virus (HIV) are eligible, if viral load is undetectable for ≥ 6 months prior to enrollment, and subjects are receiving effective anti-retroviral HIV therapy, if indicated. HIV testing is not required for subjects without a known history of HIV, unless mandated by a local health authority.
    2. For patients with a known history of HBV infection, a hepatitis B core antibody test should be conducted at screening. If positive, hepatitis B DNA testing will be performed and if active HBV infection is ruled out, the patient may be eligible.
    3. Patients who are HCV antibody positive with polymerase chain reaction negative for HCV RNA may be eligible
12. Other concurrent medical or psychiatric conditions that, in the investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
13. Received prior chemotherapy or HER2-targeted therapy for advanced or mBC.
14. Prior exposure in the adjuvant setting to an antibody-drug conjugate containing an exatecan derivative (topoisomerase I inhibitor), with a disease-free interval of less than 12 months since the last dose
15. Requirement for ongoing therapy with or prior use of any prohibited medications.
16. Participation in other studies involving investigational drug(s) within 30 days prior to enrollment or within 5 half-lives of the investigational drug(s) (whichever is longer), or participation in any other type of medical research judged not to be scientifically or medically compatible with this trial. If the patient is enrolled or planned to be enrolled in another study that does not involve an investigational drug, the agreement of the Medical Monitor is required to establish eligibility.
17. Known hypersensitivity or allergy to T-DXd, their metabolites, formulation excipient, or other monoclonal antibodies.
18. Positive serum pregnancy test or women who are lactating.
19. Only applicable in France: patients deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of T-DXd as a first-line therapy - TFST | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Time to first subsequent anti-cancer therapy (TFST) is defined as the time from the date of first dose of the study treatment to the date of i) first subsequent anti-cancer therapy after disease progression or discontinuation of maintenance treatment (in patients who discontinued due to treatment-related toxicities), or ii) death from any cause, whichever occurs first
Health-related quality of life | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdrawal of consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled.
  Time to 10% physical functioning deterioration, based on the EORTC QLQ-C30 Physical Functioning scale. Values range from 0 to 100. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Adverse events (safety) | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Occurrence /severity of AEs, laboratory abnormalities, discontinuation rates, dose reductions/interruptions
Percentage of any acute or delayed nausea and vomiting | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Percentage of any acute or delayed nausea and vomiting or breakthrough anti-emetic use, in patients receiving prophylactic anti-emetic agents (combination regimen of 3 medicinal products)
Unplanned healthcare utilization | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Composite of ER visits, unplanned hospitalizations and non-programed visits
Efficacy of T-DXd as a first-line therapy - PFS | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Progression-free survival, defined as the time from the date of first dose to the date of first clinical or radiological progression or death due to any cause, whichever occurs first, as assessed by the investigators' assessments and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Efficacy of T-DXd as a first-line therapy - ORR | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Overall response rate (ORR), defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) as per local investigator's assessment and according to RECIST 1.1
Efficacy of T-DXd as a first-line therapy - CBR | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Clinical benefit rate (CBR), defined as the proportion of patients with a best overall response of i) CR or PR or ii) SD or Non-CR/Non-PD lasting more than 24 weeks as per local investigator's assessment and according to RECIST 1.1
Efficacy of T-DXd as a first-line therapy - TtR | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Time to response (TtR), defined as the time from the date of first dose to the first objective tumor response (tumor shrinkage of ≥30%) observed for patients who achieved a CR or PR
Efficacy of T-DXd as a first-line therapy - DoR | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Duration of response (DoR), defined as the time from the first occurrence of a documented objective response (CR or PR) to disease progression, as per local investigator's assessment and according to RECIST 1.1., or death from any cause, whichever occurs first
Patient reported outcomes for HrQoL - EORTC QLQ-C30 | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  1. Proportion of participants experiencing treatment-related symptoms as measured by selected scales from the EORTC QLQ-C30 - higher scores are associated with greater symptom severity.
  2. Change from baseline in the global health status (GHS)/QoL scale - higher score means better overall health;
  3. Time to 10% deterioration in the GHS/QoL scale - higher scores mean a better outcome
Patient reported outcomes for HrQoL - EORTC QLQ-BR42 | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Proportion of participants experiencing treatment-related symptoms as measured by selected scales from the EORTC QLQ-BR42 - higher scores are associated with greater symptom severity.
Patient reported outcomes for HrQoL - CTCAE | Day 1 of each cycle until Cycle 9 (each cycle is 21 days)
  Proportion of participants with maintained or improved treatment-related self-reported symptoms.
Digital health tools - Adherence | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  The study will also evaluate digital health adherence and utilization and identify factors predictive of digital health adherence. Usage patterns in digital health interventions vary (e.g., no use, partial use, early discontinuation, or full adherence). Adherence, defined by Donkin et al. as "the degree to which the user followed the program as designed," (Donkin et al. 2011) is generally linked to greater effectiveness, though alternative patterns may still meet treatment goals. Evaluating adherence and predictors of usage in cancer care is essential to improve design, tailoring, and engagement. In this study, patients will be group based on their digital adherence. This grouping will be performed by dividing the overall study population into tertiles according to their cumulative digital usage data. The groups will represent low, medium, and high digital adherence.
Digital health tools - Patient typology and software solutions | From date of enrollment until the date of first documented progression, death, lost of follow-up, withdraw consent or the study is terminated by SOLTI, whichever occurs first, assessed up to approximately 60 months after the first patient enrolled
  Comparative descriptive studies of outcome factors (e.g. patient reported outcomes, efficacy, adherence) in subgroups defined by individual patient characteristics, population, and software solution.

CONTACTS AND LOCATIONS:
Locations (3):
- Gustave Roussy, Villejuif, France
- Klinikum der Universitaet Muenchen AöR, München, Germany
- Hospital Universitari Vall d'Hebrón, Barcelona, Barcelona, Spain